CLINICAL TRIAL: NCT01441830
Title: Treatment of Subacromial Shoulder Pain
Brief Title: Radial Extracorporeal Shock Wave Therapy (rESWT) Treatment of Subacromial Shoulder Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011/5347
Record Dates: First submitted 2011-09-15; First posted 2011-09-28 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Shoulder Impingement Syndrome; Subacromial Shoulder Pain
Keywords: shoulder; subacromial; impingement; tendinopathy; rESWT; shock wave; ESWT; RSWT
MeSH Terms: conditions — Shoulder Impingement Syndrome; Tendinopathy | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sham rESWT (Sham Comparator)
  Interventions: Device: Radial extracorporeal shock wave therapy
- rESWT (Active Comparator)
  Interventions: Device: Radial extracorporeal shock wave therapy

INTERVENTIONS:
Device: Radial extracorporeal shock wave therapy — The shockwave treatment will be administered once a week for four weeks on one to three specific points (supraspinatus, infraspinatus or subscapular tendon)and with a pressure between 1,5-3 Bar
  Other Names: rESWT; ESWT; RSWT; shock wave therapy

SUMMARY:
The purpose of this study is to determine whether rESWT (radial extracorporeal shock wave therapy) combined with supervised exercises will improve function and reduce pain in subacromial shoulder pain compared with supervised exercises alone.

ELIGIBILITY:
Inclusion Criteria:

* Dysfunction or pain on abduction
* Pain on one of two isometric tests (abduction or external rotation)
* Positive Hawkins sign
* Normal passive glenohumeral range of motion

Exclusion Criteria:

* Previous surgery on affected shoulder
* Instability
* Total rupture of the rotator cuff (evaluated clinically or by US)
* Clinical signs of a cervical syndrome
* Infection in the area
* Exclusion criteria cont.
* Patients considered unable to fill out questionnaires or to go through the treatment
* Use of anticoagulant drugs or bleeding disorder
* Pregnancy
* Previous experience of one of the study interventions
* Corticosteroid injection in the past 6 weeks.
* SPADI < 20

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 24 weeks

SECONDARY OUTCOMES:
Health-related quality of life (Eq-5d) | 24 weeks and 1 year
Return to work | 6 weeks, 12 weeks, 24 weeks and 1 year
Pain and function measured on a 11 point Likert type scale | 6 weeks, 12 weeks, 24 weeks and 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Ulleval, department for physical medicine and rehabilitation, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Kvalvaag E, Anvar M, Karlberg AC, Brox JI, Engebretsen KB, Soberg HL, Juel NG, Bautz-Holter E, Sandvik L, Roe C. Shoulder MRI features with clinical correlations in subacromial pain syndrome: a cross-sectional and prognostic study. BMC Musculoskelet Disord. 2017 Nov 21;18(1):469. doi: 10.1186/s12891-017-1827-3. PMID 29157224
- [Derived] Kvalvaag E, Brox JI, Engebretsen KB, Soberg HL, Juel NG, Bautz-Holter E, Sandvik L, Roe C. Effectiveness of Radial Extracorporeal Shock Wave Therapy (rESWT) When Combined With Supervised Exercises in Patients With Subacromial Shoulder Pain: A Double-Masked, Randomized, Sham-Controlled Trial. Am J Sports Med. 2017 Sep;45(11):2547-2554. doi: 10.1177/0363546517707505. Epub 2017 Jun 6. PMID 28586628
- [Derived] Kvalvaag E, Brox JI, Engebretsen KB, Soberg HL, Bautz-Holter E, Roe C. Is radial Extracorporeal Shock Wave Therapy (rEWST) combined with supervised exercises (SE) more effective than sham rESWT and SE in patients with subacromial shoulder pain? Study protocol for a double-blind randomised, sham-controlled trial. BMC Musculoskelet Disord. 2015 Sep 11;16:248. doi: 10.1186/s12891-015-0712-1. PMID 26361756